CLINICAL TRIAL: NCT04181021
Title: Evaluation of Values Clarification and Attitude Transformation Workshops on Abortion and Family Planning Service Provision and Client Experience in Socially Franchised Facilities in Ethiopia: A Cluster Randomized Study
Brief Title: Evaluation of Values Clarification and Attitude Transformation Workshops on Abortion and Family Planning Service Provision and Client Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibis Reproductive Health (Other)
Collaborators: Marie Stopes International (Other); Marie Stopes Ethiopia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019VCAT
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Abortion; Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Providers and community-based promoters will participate in the VCAT workshop. Providers and community-based promoters will take part in two different workshops at different times.
  Interventions: Behavioral: Values Clarification and Attitudes Transformation (VCAT) Workshop
- Control (No Intervention): Providers and promoters in the control arm will not be invited to participate in the VCAT workshop.

INTERVENTIONS:
Behavioral: Values Clarification and Attitudes Transformation (VCAT) Workshop — VCAT is a participatory workshop aimed to provide accurate information about abortion and family planning and space to engage in critical self-reflection, provoke dialogue on beliefs, values and professional ethics and responsibilities around providing abortion and contraceptive care, and provide a deeper understanding of the range of circumstances in which women seek abortion and contraception.
  Arms: Intervention

SUMMARY:
Stigma around abortion and other reproductive health care is pervasive in most contexts and has been documented to have implications for the quality of care. This study aims to assess how Values Clarification and Attitude Transformation (VCAT) workshops for providers of abortion and family planning services influences service provision of abortion and family planning services, including the quality and person-centeredness of care provided. A secondary aim is to measure how provider attitudes, knowledge, and behavioral intent change over time as a result of the VCAT workshop.This study will be conducted across multiple regions in Ethiopia.

DETAILED DESCRIPTION:
This two-arm, parallel design stratified cluster randomized control trial aims to assess how Values Clarification and Attitude Transformation (VCAT) workshops on influences service provision to clients seeking abortion and family planning services. The study aims to assess whether the experiences and quality of care of abortion clients of any age and family planning clients under the age of 20 change as a potential consequence of the VCAT workshop. A secondary aim is to measure how provider attitudes, knowledge, and behavioral intent change over time in relation to the VCAT workshops. This study will be conducted at socially franchised facilities in the Blue Star network in Ethiopia run by Marie Stopes Ethiopia. This study is a mixed methods study with two concurrent quantitative study designs that account for the need for different recruitment and data collection strategies for the two target populations, clients and providers, and a qualitative component for both target populations.

The unit of randomization is the facility. Facilities will be randomized with a 1:1 ratio between intervention and control within strata defined by eligible client volume, using a disproportionate allocation by client volume. Facilities will not be blinded to treatment assignment group after baseline. To measure client experience of person-centered quality care, cross-sectional surveys with adolescent clients under 20 years old who receive family planning or abortion services, and with abortion clients of any age will be collected at two time points (before and after VCAT workshops). Clients will only be recruited from "high" volume facilities. Providers and promoters will be followed longitudinally for up to 6 months. A subsample of abortion clients who participated in the survey will be interviewed. Using preliminary analysis of provider responses, semi-structured in-depth interviews (IDI) with a subset of providers who took part in the VCAT training will be conducted. Providers from facilities who demonstrated significant change in outcomes of interest and those who did not will be purposively sample.

Additionally, service volume and referrals of abortion and family planning clients will be analyzed for all facilities using routine service statistics to assess whether there was a potential change in volumes related to the VCAT workshops.

ELIGIBILITY:
Eligibility Criteria for clients:

* Be willing to participate
* Speak a language that is spoken by a study staff member
* Be able to give informed consent
* Have obtained abortion services (any age) or family planning services (<20 years old) from one of the participating social franchise facilities during one of the study periods

Eligibility Criteria for providers:

* Be trained to provide medication abortion and/or surgical abortion or be a community-based promoter employed by participating Blue Star facilities
* Speak one of the study languages, including English, Amharic, Oromiffa, and Tigrinya.
* Be willing to be randomized to either participate in VCAT training or be in the control arm.
* Be willing to participate in the study
* Be able to provide informed consent
* Have a private space in the clinic for clients to complete the client survey and in-depth interview
* Not have participated in 2018 pilot VCAT trainings
* Work at a facility that has been a part of the social franchise network for at least six months prior to the study

Eligibility criteria for promoters

* Speak a language spoken by a study staff member
* Be willing to participate in the study
* Be willing to be randomized to participate in the VCAT training for community-based promoters

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Person-centered abortion and family planning scale | 1.5 months
  A validated scale measuring the dimensions of respectful and supportive care, communication and autonomy, and structural quality. The score is on a scale from 0 to 69 and higher scores represent more person-centered care.
Percent of clients reporting essential person-centered care components | 1.5 months
  Percent of clients reporting having received kind and compassionate care from their provider, not feeling like they were treated differently based on age, marital status, or other characteristic, not feeling judged by their provider, having received respectful care, and feeling involved in the decisions around their care

SECONDARY OUTCOMES:
Percent of providers that agree they could support a woman having an abortion or using family planning if they didn't agree with their decision | 6 months
  Agreement with the following four measures that capture agreement with providing abortion and family planning even in cases where providers may have conflicted values: I feel comfortable performing a safe abortion procedure for anyone who requests it regardless of the reason,I support a client's decision to have a safe abortion even if I didn't agree with her decision, I could provide family planning to a client even if I thought they were too young to be using contraception, I feel comfortable removing IUDs or implants even if I think the client shouldn't have it removed
Level of knowledge around interpretation for legal grounds for abortion in Ethiopia | 6 months
  Proportion knowing the legal indications for abortion in Ethiopia, the legal grounds for denial of abortion services, and the correct interpretation of the law around abortion services for married women, minors, women seeking services under the rape and incest clause, and women requesting an abortion under the grounds that the pregnancy is a risk to their health
Volume of patients | 1 year
  Volume of abortion and family planning clients under age 20
Patient referrals by promoters | 1 year
  Number of referrals for safe abortion care and for family planning among clients under the age of 20
Percent of providers who believe that women should have access to safe, comprehensive abortion care regardless of COVID-19 in Ethiopia | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Wollum, Principal Investigator — Ibis Reproductive Health
Locations (1):
- Blue Star facilities, Multiple, Addis Ababa, Oromiya, Tigray, Snnpr, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wollum A, Key K, Mersha T, Nicholson M, Page G, Austen K, Endale ME, Moseson H. Does a values clarification and attitudes transformation (VCAT) workshop influence provider attitudes, knowledge, and service provision related to abortion care?: Evidence from a mixed-methods longitudinal randomised controlled trial in Ethiopia. Glob Public Health. 2025 Dec;20(1):2465643. doi: 10.1080/17441692.2025.2465643. Epub 2025 Feb 21. PMID 39984306